CLINICAL TRIAL: NCT03651739
Title: Knee Connect: Measuring Range of Motion and Gait Metrics After Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 02KINERIS2017
Record Dates: First submitted 2018-08-09; First posted 2018-08-29 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Rehabilitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- TKR Patients: Any patient undergoing total knee arthroplasty and will use the Knee Connect during their knee classes at the Holland Centre
  Interventions: Device: Knee Connect

INTERVENTIONS:
Device: Knee Connect — An electronic goniometer with smart phone application

SUMMARY:
The main goals of total knee replacement (TKR) surgery are to relieve pain and to allow patients to remain active. Sunnybrook is working with Kineris Inc.to advance a wearable device, the Knee Connect, aimed at tracking the physical recovery of patients after total knee replacements. After surgery, patients experience a gradual progression in function as their knee range of motion (ROM) increases and their gait patterns normalize. Goals for these metrics are well documented after the patient is fully recovered. However, there is a lack of detailed information available about the week by week improvements patients make in these metrics. The main objective of this study is to determine the accuracy of the Knee Connect device in quantifying the weekly improvements in ROM and gait parameters of patients recovering from surgery.

DETAILED DESCRIPTION:
A research assistant will conduct in person data collections on 36 patients using the Kineris wearable device. The device is an electronic goniometer connected to a smart phone application. Patients will be recruited from the "Patient Orientation Program" (POP) at the Sunnybrook Holland Centre. Data collection will occur preoperatively, at the end of each physiotherapy Knee Class session, and at the three month postoperative clinic visit. The research assistant will help fit and attach the wearable device to each patient's knee. Patients will be asked to bend their knee (flexion and extension) while wearing the device which will measure patients range of motion. The research assistant will also measure knee range of motion using a handheld protractor. Afterward, patients will be asked to walk 10 steps, using any walking aids or techniques they typically use at home. There will be 15 collections per patient requiring ten minutes per session. Chart reviews will also be conducted to determine patient reported outcomes which will be then correlated with the functional measures.

All data will be extracted and input into an excel file. For both the ROM tests, the accuracy of the Knee Connect device will be compared against the plastic goniometer. This will be done by using a paired t-test and calculating interclass correlation coefficient. The data will then be analyzed using a repeated measures ANOVA and Bonferroni post-hoc analysis to determine differences in the variables week to week. Additionally, a regression analysis will be used to estimate the week by week improvements in these variables.

ELIGIBILITY:
Inclusion Criteria:

* Be currently on the waiting list for a primary TKR
* Be enrolled for the "Knee Class" postoperative physiotherapy at the Sunnybrook Holland Centre with the expectation of attending the class through the duration of the class.
* Be able to provide informed consent.

Exclusion Criteria:

* Revision total knee arthroplasty
* Neuromuscular disorder
* Bilateral TKR procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from the Patient Orientation Program clinic, approximately 4-6 weeks pre-surgery. Patients must be available for testing at the end of every Knee Class therapy session, for the duration of their Knee Class visits.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Knee Range of Motion Error | One reading 2-4 weeks pre-operation, two readings weekly for 2-6 weeks post-operation (during physiotherapy knee class visits), one during 3 month post-operative clinic visit
  The difference in measured knee range of motion (in degrees) between the Knee Connect and the handheld goniometer.
  Completed at each study time point (listed below) in order to gather as much data on the accuracy of knee connect compared to the goniometer.

SECONDARY OUTCOMES:
Knee range of motion | One reading 2-4 weeks pre-operation, two readings weekly for 2-6 weeks post-operation (during physiotherapy knee class visits), one during 3 month post-operative clinic visit
  The weekly knee range of motion (in degrees) measured by the Knee Connect
Stride Time | One reading 2-4 weeks pre-operation, two readings weekly for 2-6 weeks post-operation (during physiotherapy knee class visits), one during 3 month post-operative clinic visit
  The weekly gait stride time (in seconds) measured by the Knee Connect
Stance Range of Motion | One pre-operative, one during inpatient stay, 12 during knee class visits, one during 3 month clinic visit
  The weekly gait stance range of motion (in degrees) measured by the Knee Connect
Swing Range of Motion | One reading 2-4 weeks pre-operation, two readings weekly for 2-6 weeks post-operation (during physiotherapy knee class visits), one during 3 month post-operative clinic visit
  The weekly gait swing range of motion (in degrees) measured by the Knee Connect
Western Ontario and McMaster Universities Osteoarthritis Index | One at 6 week visit, one during 3 month clinic visit
  Western Ontario and McMaster Universities Osteoarthritis Index function sub-scale and total score
  Sub scales: Pain (5 items, each rated on a scale from 0-4); Joint stiffness (2 items, each rated on a scale from 0-4), Physical function (17 items, each rated on a scale from 0-4 for level of difficulty)
  Score range: Pain subscale 0-20 WOMAC points; Joint stiffness subscale 0-8 WOMAC points. Physical function subscale 0-68 WOMAC points. Total score 0-96 WOMAC points (96 = worse pain, stiffness and physical function). Subscales are summed for total score

CONTACTS AND LOCATIONS:
Overall Officials: David Wasserstein, MD, Principal Investigator — Sunnybrook Hospital
Locations (1):
- Sunnybrook Holland Orthopaedic & Arthritic Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chiang CY, Chen KH, Liu KC, Hsu SJ, Chan CT. Data Collection and Analysis Using Wearable Sensors for Monitoring Knee Range of Motion after Total Knee Arthroplasty. Sensors (Basel). 2017 Feb 22;17(2):418. doi: 10.3390/s17020418. PMID 28241434
- [Background] Dennis DA, Komistek RD, Stiehl JB, Walker SA, Dennis KN. Range of motion after total knee arthroplasty: the effect of implant design and weight-bearing conditions. J Arthroplasty. 1998 Oct;13(7):748-52. doi: 10.1016/s0883-5403(98)90025-0. PMID 9802659
- [Background] Steiner ME, Simon SR, Pisciotta JC. Early changes in gait and maximum knee torque following knee arthroplasty. Clin Orthop Relat Res. 1989 Jan;(238):174-82. PMID 2910598
- [Background] Chao EY, Laughman RK, Stauffer RN. Biomechanical gait evaluation of pre and postoperative total knee replacement patients. Arch Orthop Trauma Surg (1978). 1980;97(4):309-17. doi: 10.1007/BF00380714. PMID 7458617
- [Background] Wilson SA, McCann PD, Gotlin RS, Ramakrishnan HK, Wootten ME, Insall JN. Comprehensive gait analysis in posterior-stabilized knee arthroplasty. J Arthroplasty. 1996 Jun;11(4):359-67. doi: 10.1016/s0883-5403(96)80023-4. PMID 8792240
- [Background] Seel T, Raisch J, Schauer T. IMU-based joint angle measurement for gait analysis. Sensors (Basel). 2014 Apr 16;14(4):6891-909. doi: 10.3390/s140406891. PMID 24743160
- [Background] Mizner RL, Petterson SC, Clements KE, Zeni JA Jr, Irrgang JJ, Snyder-Mackler L. Measuring functional improvement after total knee arthroplasty requires both performance-based and patient-report assessments: a longitudinal analysis of outcomes. J Arthroplasty. 2011 Aug;26(5):728-37. doi: 10.1016/j.arth.2010.06.004. Epub 2010 Sep 20. PMID 20851566